CLINICAL TRIAL: NCT05625035
Title: Efficacy and Safety of Lianhua Qingwen in the Long-Term Rehabilitation of Patients With Coronavirus Infection: a Randomized, Open-Label, Comparative Study
Brief Title: Lianhua Qingwen for the Rehabilitation of Patient With Coronavirus Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lianhua Qingwen 2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Coronavirus; Traditional Chinese Medicine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lianhua Qingwen plus conventional therapy (Experimental)
  Interventions: Drug: Lianhua Qingwen capsules
- Conventional therapy (No Intervention)

INTERVENTIONS:
Drug: Lianhua Qingwen capsules — Lianhua Qingwen capsules: 4 capsules once, three times daily
  Arms: Lianhua Qingwen plus conventional therapy

SUMMARY:
The patients with coronavirus infection usually have fever, respiratory symptoms, headache, toothache, muscle soreness, physical decline, and so on, while others are asymptomatic patients. It is urgent to find drugs to improve the long-term rehabilitation of symptomatic patients with coronavirus infection and decrease the duration of viral shedding in both symptomatic and asymptomatic patients. This study aims to investigate the efficacy and safety of Lianhua Qingwen capsules in patients with coronavirus infection. The duration of viral shedding and symptoms before discharge, as well as the negative conversion ratio and disappearance ratio of main symptoms after 7-day treatment, will be evaluated. 6-month follow-up will be performed to evaluate the effect of Lianhua Qingwen on all infection events and the long-term rehabilitation of the symptoms induced by coronavirus infection.

ELIGIBILITY:
Inclusion Criteria:

* confirmed SARS-CoV-2 Infection by virus testing;
* ≥18 years of age;
* informed consent provided.

Exclusion Criteria:

* overt bacterial infection in the respiratory tract resulting from common pathologies, including primary immunodeficiency disease, acquired immunodeficiency syndrome, congenital respiratory malformation, congenital heart disease, gastroesophageal reflux disease, and abnormal lung development;
* asthma treated daily, chronic airway disease, respiratory bacterial infections (e.g., purulent tonsillitis), acute tracheobronchitis, sinusitis, otitis media, and further respiratory tract pathologies potentially affecting the trial's data analysis;
* common pulmonary diseases (e.g., severe pulmonary interstitial lesions and bronchiectasis) confirmed by chest CT;
* severe pneumonia requiring ventilator use;
* previous or present diseases potentially affecting trial participation or influencing study outcome, based on the investigator's judgment;
* pregnancy or lactation in women;
* participation in a clinical study in the past 3 months;
* history of allergy to ≥2 drugs or foods or known allergy to the drug's constituents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all Infection events | From discharge to 6 months
  Recurrence coronavirus infection or any new infection events

SECONDARY OUTCOMES:
Duration of viral shedding | 6 months
Negative conversion ratio | 7 days
Positive conversion ratio | From discharge to 6 months
Duration of main symptoms before discharge | 6 months
Disappearance ratio of main symptoms | 7 days
Recurrence frequency of main clinical symptoms | From discharge to 6 months
Mean duration of main clinical symptoms | From discharge to 6 months
Heart rate | 6 months
Heart rate | 7 days
Heart rate | Baseline
Blood pressure | 6 months
  both systolic and diastolic blood pressure
Blood pressure | 7 days
  both systolic and diastolic blood pressure
Blood pressure | Baseline
  both systolic and diastolic blood pressure
Infection events except SARS-CoV-2 | From discharge to 6 months
Frequency of fever | From discharge to 6 months
Mean duration of fever | From discharge to 6 months
Duration of fever before discharge | 6 months
Disappearance ratio of fever | 7 days
Frequency of respiratory symptoms | From discharge to 6 months
Mean duration of respiratory symptoms | From discharge to 6 months
Duration of respiratory symptoms before discharge | 6 months
Disappearance ratio of respiratory symptoms | 7 days
Frequency of nasal congestion or runny nose | From discharge to 6 months
Mean duration of nasal congestion or runny nose | From discharge to 6 months
Duration of nasal congestion or runny nose before discharge | 6 months
Disappearance ratio of nasal congestion or runny nose | 7 days
Frequency of chest distress | From discharge to 6 months
Mean duration of chest distress | From discharge to 6 months
Duration of chest distress before discharge | 6 months
Disappearance ratio of chest distress | 7 days
Frequency of palpitations | From discharge to 6 months
Mean duration of palpitations | From discharge to 6 months
Duration of palpitations before discharge | 6 months
Disappearance ratio of palpitations | 7 days
Frequency of pharyngeal discomfort | From discharge to 6 months
Mean duration of pharyngeal discomfort | From discharge to 6 months
Duration of pharyngeal discomfort before discharge | 6 months
Disappearance ratio of pharyngeal discomfort | 7 days
Frequency of headache | From discharge to 6 months
Mean duration of headache | From discharge to 6 months
Duration of headache before discharge | 6 months
Disappearance ratio of headache | 7 days
Frequency of dizziness | From discharge to 6 months
Mean duration of dizziness | From discharge to 6 months
Duration of dizziness before discharge | 6 months
Disappearance ratio of dizziness | 7 days
Frequency of toothache | From discharge to 6 months
Mean duration of toothache | From discharge to 6 months
Duration of toothache before discharge | 6 months
Disappearance ratio of toothache | 7 days
Frequency of muscle soreness | From discharge to 6 months
Mean duration of muscle soreness | From discharge to 6 months
Duration of muscle soreness before discharge | 6 months
Disappearance ratio of muscle soreness | 7 days
Frequency of physical decline | From discharge to 6 months
Mean duration of physical decline | From discharge to 6 months
Duration of physical decline before discharge | 6 months
Disappearance ratio of physical decline | 7 days
Frequency of gastrointestinal symptoms | From discharge to 6 months
Mean duration of gastrointestinal symptoms | From discharge to 6 months
Duration of gastrointestinal symptoms before discharge | 6 months
Disappearance ratio of gastrointestinal symptoms | 7 days
Frequency of urinary symptoms | From discharge to 6 months
Mean duration of urinary symptoms | From discharge to 6 months
Duration of urinary symptoms before discharge | 6 months
Disappearance ratio of urinary symptoms | 7 days
Drug-related adverse events | 6 months
Drug-related adverse events | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Panpan Hao, MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- International Convention and Exhibition Center Shelter Hospital, Ürümqi, Xinjiang, China